CLINICAL TRIAL: NCT05558254
Title: Feasibility and Effect Size of an Intervention to Enhance Muscle Strength Assisted by Robotic Technology (ROBERT®) in Subacute Rehabilitation After Spinal Cord Injury
Brief Title: ROBERT® as an Intervention to Enhance Muscle Strength After Spinal Cord Injury
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spinal Cord Injury Centre of Western Denmark (Other)
Collaborators: Svend Andersen Fonden (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ROBERT
Record Dates: First submitted 2021-11-12; First posted 2022-09-28 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal cord injuries; Pilot study; robot; muscle strength
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: The patient's legs will be randomised to either training with ROBERT® or usual training (control)
Who Masked: Outcomes Assessor
Masking Description: Randomization is performed after baseline assesment. The outcomes assessor will be blinded to treatment/control group at follow-up assesment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ROBERT (Active Comparator): The intervention group will receive usual practice. As add-on, the intervention leg will receive 3-4 sets of 15-20 repetitions (30 seconds rest between each set) of muscle strength training for hip flexion with ROBERT® three times a week.
  Interventions: Other: Robert - intervention to enhance muscle strength
- Control (No Intervention): Usual practice in the control group consist of 3-5 times physiotherapy a week for 8 weeks. A session last 45 minutes. The sessions are individually adapted and can contain exercise therapy, functional training, assistive devices, electrical stimulation, hydrotherapy and tread mill training.

INTERVENTIONS:
Other: Robert - intervention to enhance muscle strength — Intervention:
  Training will be conducted with the robot ROBERT®. 3 times a week for 8 weeks the patient will conduct 60 repetitions of hip flexion of one leg. The patient is lying supine. ROBERT is attached to the patient's lower leg. The physiotherapist guides the patient's leg in hip flexion and ROBERT record the movement. The ROBERT is attached to the patient's lower leg and thereby eliminating the gravity of the leg. The physiotherapist guides the patient's leg in hip flexion and ROBERT record the movement. ROBERT is set in active or guided mode and will be individually adjusted. When practice starts the patient get visual feedback to the range of movement of the hip flexion plus the amount of repetitions conducted and persisting.
  Arms: ROBERT

SUMMARY:
Spinal cord injury (SCI) is a devastating life event with long term consequences both physically and mentally. SCI is defined as either complete or incomplete according to the International Standards of the Neurological Classification of SCI. The primary consequence of a SCI is paralysis/partial paralysis affecting the person's ability to independently functioning in everyday life e.g. in and out of bed, sit to stand and walking.

To regain the ability to transfer and walk the most important prerequisite is to rebuild as much strength as possible in the lower extremities. The optimal training paradigm to increase strength in partial paralysed muscles is unclear.

Rehabilitation robots are upcoming methods to treat sensorimotor deficits after SCI.

The rehabilitation robot ROBERT might contribute to enhance muscle strength for people with very weak strength following an incomplete SCI.

The overall objective of this Ph.D project is to investigate the feasibility and effect size of a muscle strength training intervention assisted by ROBERT® for patients with SCI and severe paresis (muscle strength 1-3 in hip flexion).

DETAILED DESCRIPTION:
SCI is a devastating life event with long term consequences both physically and mentally.

To regain the ability to transfer oneself and to walk, the most important prerequisite is to rebuild as much strength as possible in the lower extremities. The optimal training paradigm to increase strength in partial paralysed muscles is unclear. The question is whether strength is best improved by applying the principles of progressive resistance training or by focusing on high repetitions with limited resistance.

Rehabilitation robots are upcoming methods to treat sensorimotor deficits after SCI. The rationale is that the use of robotics allows adaptable support and the ability to increase therapy intensity and dose while reducing the physical burden on the therapist.

The rehabilitation robot ROBERT enables the SCI patient to conduct active or guided repetitions of specific movements in the lower extremities in the early rehabilitation phase. The hypothesis is that such use will increase muscle strength faster in the recovery process than when conducting usual physiotherapist training for people with incomplete SCI.

The objective of this PhD project is to:

1. develop and feasibility test the optimal dose, timing and outcome measures and to examine feasibility, compliance and acceptability of an intervention for lower extremities for people with subacute SCI with the rehabilitation robot ROBERT?
2. conduct a pilot with-in participant randomized controlled trail to estimate the effect size of an intervention to enhance muscle strength assisted by Robotic technology (ROBERT®) in subacute rehabilitation after spinal cord injury
3. validate accelerometer-based method to identify the supine hip flexion/extension movement and be able to differentiate it from other activity movement based on the perviosely developed algorithm.

Hypothesis:

* The patients with subacute SCI and muscle strength 1-3 in manuel muscle testing of hip flexion bilateral will be able to conduct the training with Robert.
* There is a significant increase in muscle strength (hip flexion) in the leg practicing with ROBERT® for 8 weeks compared to the other leg receiving usual training. By using ROBERT® patients with very weak muscle strength are allowed to practise repetitions with the elimination of gravity and adopted resistance and guidance in the range of movement, where they don't have the strength to perform the entire range of movement.

The knowledge gained in this study will inform the design of a future RCT study and enable a power calculation.

- The refinement of the algorithm to monitor activity will be able to differentiate hip flexion from other activities in patients with SCI

Studies:

1. Feasibility study This study will be conducted prior to the pilot with-in RCT. Consecutively, 4-8 patients admitted to Spinal Cord Injury Centre of Western Denmark (SCICWD) from November 2021 - June 2022 will be recruited. Patients with SCI (< 3 month), age ≥ 18 year and muscle strength 1 - 3 in one of the lower leg muscle groups measured by manual muscle testing will be included. Exclusion criteria: previous cerebral injury or SCI, previous damage to peripheral nervous system in lower extremities, instable fractures in thorax or lower extremities, muscle strength 0, 4 or 5, weight > 150 kg.

   The patients will conduct 4 weeks training with Robert of one leg 3 times a week.

   Muscle strength will be assessed with Handheld dynamometer (HHD) MicroFET2, (Hoggan Scientific) at baseline and after 4 week. Furthermore descriptive data of recruitment capability, resulting sample characteristics, procedures of the intervention, time consumption intervention will be evaluated. Interviews will be performed to get the patient perspective of the intervention and the acceptability.

   The study has been approved by The Danish Scientific Ethics Commission (ref. no. 1-10-72-276-21).
2. Pilot with-in participant RCT It will take place at Spinal Cord Injury Centre of Western Denmark (SCICWD) from September 2022 - December 2024. 12 consecutively patients admitted to SCICWD will be recruited. To be eligible to participate participants shall have incomplete SCI (<12 months), be age ≥ 18 year and have weakened muscle strength grade 1 - 3 in hip flexion bilateral measured by manual muscle testing due to SCI. Exclusion criteria were: Previous cerebral injury or SCI, previous damage to peripheral nervous system in lower extremities, instable fractures in thorax or lower extremities, muscle strength 0, 4 or 5 in hip flexion, weight > 150 kg.

   The patient's legs will be randomised to either training with ROBERT® or usual training (control). The Control group/leg will recieve usual practice consisting of 3-5 times physiotherapy a week for 8 weeks. A session last 45 minutes. The sessions are individually adapted and can contain exercise therapy, functional training, assistive devices, electrical stimulation, hydrotherapy and tread mill training.

   Intervention group will receive usual practice. As add-on, the intervention leg will receive 3-4 sets of 15-20 repetitions (30 seconds rest between each set) of muscle strength training for hip flexion with ROBERT® three times a week. The ROBERT is attached to the patient's lower leg and thereby eliminating the gravity of the leg. The physiotherapist guides the patient's leg in hip flexion and ROBERT record the movement. ROBERT is set in active or guided mode and will be individually adjusted. When practice starts the patient get visual feedback to the range of movement of the hip flexion plus the amount of repetitions conducted and persisting.

   From the patients' medical records the following will be collected: Age, sex, injury onset, aetiology, neurological level of injury (NLI) and American Spinal Injury Association Impairment Scale (AIS) grade, and Walking Index for SCI (WISCI). At baseline and after completing the 8 weeks intervention (2-5 days after) muscle strength will be assessed with Handheld dynamometer (HHD) (19) MicroFET2, (Hoggan Scientific) as well as electrical activity in hip flexion muscles assessed by surface Electromyography (sEMG) Keypoint, (Alpine Biomed) (20, 21) and spasticity assessed by Modified Ashworth scale (22, 23). The thickness of the rectus femoris muscle and the quadriceps femoris muscle will be assessed by ultrasound Acuson S2000 (Siemens). Number of hip flexions and activity level will be monitored with accelerometer in both legs all day for three days at baseline, at week 4 of the intervention and the week after completing the intervention.

   Parametric analyses of paired data (post-pre). Discrete variables will be examined with non-parametric analysis. Preliminary data from the feasibility study estimate that it will be realistic to enroll 8-12 persons to complete the study in the period from August 2022 till December 2023.

   The study has been approved by The Danish Scientific Ethics Commission (ref. no. 1-10-72-108-22). The study will be conducted in accordance with the Helsinki Declaration of 2008, the General Data Protection Regulation and legislation and the Data Protection Act. The study is registered at the internal list of research projects at the Central Denmark Region (Ref.nr.1-16-02-276-22).
3. Validation study This study will be conducted from May 2022-December 2022. 10 healthy adults and 10 patients with SCI admitted SCICWD will be recruited. Accelerometer will be placed with non-allergenic tape at the front and the lateral side of the test person's legs. The test persons will perform supine hip flexion/extension with and without ROBERT® as well as sit-to stand, standing, walking, cycling (Motomed) and transfer from wheelchair to bench. These movements will be recorded with accelerometer as well as video. Validation of the algorithm will be established using video recordings as gold standard.

ELIGIBILITY:
Inclusion Criteria:

* SCI (< 12 month),
* Age ≥ 18 year
* Muscle strength 1 - 3 in hip flexion in both legs measured by manual muscle testing.
* Sufficient Danish or English to be able to provide informed consent

Exclusion Criteria:

* Previous cerebral injury or SCI
* Previous damage to peripheral nervous system in lower extremities
* Instable fractures in thorax or lower extremities
* Muscle strength 0, 4 or 5 in hip flexion
* Weight > 150 kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Muscle strength in Newton | At baseline and at 8 weeks
  Change in maximal voluntary contraction (MVC) in isometric muscle strength (N) of hip flexion (8 weeks - baseline)

SECONDARY OUTCOMES:
Chance in EMG activity | At baseline and at 8 weeks
  Change in amplitude and Root Mean Square (8 weeks - baseline) of m. rectus femoris.
Change in repetitions | At baseline and at 8 weeks
  Change in number of repetitions of hip flexions in both legs (8 weeks - baseline) monitored over 3 days
Difference between legs in numbers of hip flexion | At 4 weeks
  Difference between legs in number of repetitions of hip flexions at week 4 (Intervention leg - control leg) monitored over 3 days
Change in spasticity | At baseline and at 8 weeks
  Change in spasticity in hip flexors at (8 weeks - baseline)
Change in muscle thickness | At baseline and at 8 weeks
  Change in muscle thickness rectus femoris and quadriceps femoris at (8 weeks - baseline)
Self-rated hip strength | At 8 weeks
  Difference between legs in self-rated hip strength at 8 weeks
Self-rated ability to use leg in function | At 8 weeks
  Difference between legs in self-rated ability to use the leg in function at 8 weeks

OTHER OUTCOMES:
Acceptability and suitability of the intervention - patients' perspective | At 8 weeks
  Qualitative interviews: What are patients' experiences of the intervention? Interviews will be transcribed and analysed. Emerging themes will be discussed and if possible incorporated in the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Lillelund, MSc, PT, Principal Investigator — Spinal Cord Injury Centre of Western Denmark
Locations (1):
- Spinal Cord Injury Centre of Western Denmark, Viborg, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sorensen SL, Poulsen I. Patients' and physiotherapists' experiences with robotic technologies for lower extremity rehabilitation following spinal cord injury: a reflexive thematic analysis. Disabil Rehabil. 2025 Oct 17:1-14. doi: 10.1080/09638288.2025.2573170. Online ahead of print. PMID 41105483
- [Derived] Lillelund Sorensen S, Lipperts M, Nielsen JF, Naess-Schmidt E. Clinical validation of a rule-based decision tree algorithm for classifying hip movements in people with spinal cord injury. J Spinal Cord Med. 2025 Mar 31:1-10. doi: 10.1080/10790268.2025.2472096. Online ahead of print. PMID 40163036
- [Derived] Sorensen SL, Poulsen I, Harvey LA, Biering-Sorensen F, Nielsen JF. Robotic technology (ROBERT(R)) to enhance muscle strength in the hip flexor muscles following spinal cord injury: a feasibility study. Spinal Cord Ser Cases. 2024 Apr 10;10(1):20. doi: 10.1038/s41394-024-00630-9. PMID 38600074